CLINICAL TRIAL: NCT03018288
Title: A Randomized, Double Blind Phase II Trial of Surgery, Radiation Therapy Plus Temozolomide and Pembrolizumab With and Without HSPPC-96 in Newly Diagnosed Glioblastoma (GBM)
Brief Title: Radiation Therapy Plus Temozolomide and Pembrolizumab With and Without HSPPC-96 in Newly Diagnosed Glioblastoma (GBM)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed early due to poor accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 170034; 17-C-0034
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2024-02-28 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma
Keywords: Malignant Gliomas; Immunotherapy
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — pembrolizumab; vitespin; Temozolomide; Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1/Temozolomide + Pembrolizumab + Radiation Therapy (Other): Standard treatment with experimental treatment (pembro) added.
  Interventions: Drug: Pembrolizumab; Drug: Temozolomide; Procedure: Surgery
- 2/Temozolomide+Pembrolizumab (Experimental): Temozolomide+Pembrolizumab
  Interventions: Drug: Pembrolizumab; Drug: Temozolomide; Procedure: Surgery
- 3/Temozolomide+Pembrolizumab+ Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine (Experimental): Temozolomide+Pembrolizumab+ HSPPC96 Vaccine
  Interventions: Drug: Pembrolizumab; Biological: HSPPC-96; Drug: Temozolomide
- 4/Temozolomide+Pembrolizumab+ Placebo (Placebo Comparator): Temozolomide+Pembrolizumab+ Placebo
  Interventions: Drug: Pembrolizumab; Drug: Temozolomide; Other: Placebo

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab at 200mg will be administered on day 1 as a 30-minute intravenous (IV) infusion (prior to radiation therapy (RT) every 3 weeks during RT on days 1, 22 and 43. At one year, if participants are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with heat shock protein peptide complex -96 (HSPPC 96) or placebo vaccine if any is available.
  Other Names: Keytruda
Biological: HSPPC-96 — One week post RT, patients will receive weekly x 4 a dose of heat shock protein peptide complex -96 (HSPPC 96) 0.4mL intradermal vaccine or placebo. HSPPC-96 vaccine or placebo will then be given 21 days after the day 5 dose of temozolomide (TMZ). HSPPC-96 vaccine or placebo vaccine will be given for 6 cycles or until supply runs out. Participants who receive placebo will be matched for number of vaccine injections that were generated by their tumor tissue. At one year, if participants are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with HSPPC-96 or placebo vaccine if any is available.
  Other Names: heat shock protein peptide complex -96 (HSPPC 96)
  Arms: 3/Temozolomide+Pembrolizumab+ Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine
Drug: Temozolomide — Temozolomide (TMZ) will be administered on day 1 of radiation therapy (before radiation therapy (RT) treatment) and continue throughout RT at the dose of 75 mg/m^2. Post RT: The starting TMZ dose will be 150 mg/m^2/day for cycle 1, days 1-5, with a single dose escalation to 200 mg/m^2/day (days 29-33) and for all subsequent treatment if no treatment-related adverse events greater than Grade 2 are noted. TMZ will be given for 6 cycles.
  Other Names: Temodar
Other: Placebo — One week post radiation therapy (RT), participants will receive weekly x 4 a dose of heat shock protein peptide complex -96 (HSPPC 96) 0.4mL intradermal vaccine or placebo. HSPPC-96 vaccine or placebo will then be given 21 days after the day 5 dose of Temozolomide (TMZ). HSPPC-96 vaccine or placebo vaccine will be given for 6 cycles or until supply runs out. Participants who receive placebo will be matched for number of vaccine injections that were generated by their tumor tissue. At one year, if participants are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with HSPPC-96 or placebo vaccine if any is available.
  Arms: 4/Temozolomide+Pembrolizumab+ Placebo
Procedure: Surgery — Tissue for vaccine production and neo-epitope monitoring.
  Arms: 1/Temozolomide + Pembrolizumab + Radiation Therapy; 2/Temozolomide+Pembrolizumab

SUMMARY:
Background:

Glioblastoma (GBM) refers to a specific kind of brain cancer called glioblastoma. The standard treatment for GBM is radiation plus temozolomide, an oral chemotherapy drug. Pembrolizumab is an immune therapy that is now used to treat other cancers. The addition of pembrolizumab to the standard treatment of radiation and temozolomide has been shown to be well tolerated. Researchers want to see if adding a vaccine made from the person's own tumor will improve the effect of the pembrolizumab. The vaccine which is developed from fresh tumor taken at the time of surgery is called heat shock protein peptide complex-96 (HSPPC-96).

Objectives:

To see if the adding of pembrolizumab and HSPPC-96 improves the standard treatment for glioblastoma.

Eligibility:

Adults at least 18 years old with glioblastoma.

Design:

Participants will be screened with typical cancer tests:

Brain scan

Medical history

Blood and urine tests

Questions about quality of life and symptoms

These tests will be repeated throughout the study.

Participants will have surgery to remove their tumor. A tissue sample from the tumor will be sent to a lab. A vaccine will be made from it.

Some participants will get pembrolizumab and vaccine. Some will get pembrolizumab and placebo. Participants will not know which they get.

Participants will get radiation for 6 weeks.

Participants will take temozolomide by mouth before each treatment.

Participants will get pembrolizumab by intravenous (IV) for 30 minutes 3 times over the radiation cycle.

Participants will keep taking the 2 drugs every few weeks for about a year. Some may take pembrolizumab for an additional year.

Most participants will get the vaccine or placebo after radiation. They will get it 5 times over 6 weeks. Some participants will continue to get the vaccine every few weeks for 1 or 2 years.

Participants will repeat the screening tests when they stop study treatment. They will also have follow-up phone calls.

DETAILED DESCRIPTION:
Background:

* Malignant gliomas are unfortunately, in most cases, a uniformly fatal tumor. Despite aggressive surgery, radiation treatment (RT) and chemotherapy at initial diagnosis these tumors almost always recur.
* Many clinical trials in glioblastoma (GBM) have evaluated the addition of agent(s) to standard therapy which consists of concurrent radiation with temozolomide chemotherapy after maximal surgical resection in patients with newly diagnosed disease and salvage chemotherapy with either rechallenge with temozolomide or an alternative alkylating agent such as lomustine (CCNU) or cisplatin. To date, none of the combination strategies have demonstrated clinical benefit. Furthermore, in subjects with an unmethylated MGMT (O6-methylguanine-DNA methyltransferase) promoter temozolomide has only modest benefit and salvage therapies have not demonstrated a significant impact in this subject group underscoring the need for more research.
* Immunotherapy offers the promise of improving outcomes for patients with GBM by evoking specific immune responses that may produce a more sustained and less toxic effect than conventional therapy. Heat-shock proteins (HSPs), which function as intracellular chaperones, can be used to deliver a variety of tumor antigens to antigen presenting cells for immune stimulation.
* Heat Shock Protein-Peptide Complex-96 (HSPPC-96) consists of the heat shock protein glycoprotein-96 (HSP gp-96) and a wide array of chaperoned proteins, including autologous antigenic peptides (aka vaccine). Heat shock proteins (HSP) are molecules that respond to cellular stress and counteract abnormal protein folding. They are known to modulate immune responses, especially the HSP gp-96. In a stressful environment, such as a tumor, HSPs are upregulated and highly expressed on tumor cells. This protects the tumor and leads to resistance to therapy. HSP expression is associated with cellular proliferation, apoptosis evasion, tissue invasion, metastasis, and angiogenesis.
* Pembrolizumab is a potent and highly selective humanized monoclonal antibody (mAb) of the immunoglobulin G4 (IgG4)/kappa isotype designed to directly block the interaction between Programmed cell death protein 1 (PD-1) and its ligands, programmed death-ligand 1 (PD-L1) and programmed cell death-ligand 2 (PD-L2). Additionally, pembrolizumab is thought to also have activity in the peripherally circulating T-effector cells by reversing lymphocyte exhaustion. It is currently Food and Drug Administration (FDA) approved for use in patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor and non-small cell lung cancer (NSCLC) with elevated PD-L1 in the tumor. recurrent or metastatic HNSCC with disease progression on or after platinum-containing chemotherapy. It is also FDA approved for use with advanced (metastatic) non-small cell lung cancer (NSCLC) whose disease has progressed after other treatments and with tumors that express a protein called PD-L1 and for the treatment of patients with recurrent or metastatic head and neck squamous cell carcinoma (HNSCC) with disease progression on or after platinum-containing chemotherapy.
* This study will be the first to evaluate this combination of vaccine (HSPPC-96) and PD-1 inhibition (pembrolizumab) in newly diagnosed GBM patients whose tumors are MGMT promoter unmethylated and are isocytrate dehydrogenase (IDH) wildtype; and will provide important data on immune-modulatory effect of this combination. This may be of particular value in patients with high peripheral PD-L1 expression, but also the value of PD-1 added to standard GBM therapy. As vaccine needs to be generated from the patient s tumor, patients will need to be identified prior to surgery.

Eligibility:

* MRI findings consistent with a suspected GBM or histologically confirmed newly diagnosed GBM that has not been treated and would benefit from further surgical resection.
* Tumor must be supratentorial.
* GBM diagnosis must be made by surgical excision (stereotactic biopsy will not be allowed unless there is plan for second surgery to remove greater than or equal to 80% of the tumor) and patients tumors must not have O6-Methylguanine-deoxyribonucleic acid (DNA) Methyltransferase (MGMT) promoter methylation and must be isocitrate Dehydrogenase (IDH) wildtype.
* No prior treatment with radiation or chemotherapy for their GBM.
* Age greater than or equal to 18 years on day of signing informed consent

Objective:

- The primary endpoint is to determine whether the one-year overall survival (OS) rate is improved in newly diagnosed GBM patients whose tumors have an unmethylated MGMT promoter and are IDH wildtype treated with radiation therapy (RT) + temozolomide (TMZ) + Pembrolizumab followed by TMZ + Pembrolizumab + HSPPC-96 vaccine or Placebo vaccine x 6 cycles (1 cycle is 9 weeks).

Design:

* This will be a randomized, double blind phase II trial of surgery, RT + TMZ + Pembrolizumab followed by TMZ + Pembrolizumab +/- HSPPC-96 in newly diagnosed GBM patients whose tumors have an unmethylated MGMT promoter and are IDH wildtype.
* Subjects will be assigned to intervention based on ability to generate vaccine as follows:

  * If >= 80 % of tumor removed, >=7 g of tumor is resected but HSPPC-96 cannot be generated, subjects will be treated on the ancillary arm of RT+TMZ +Pembrolizumab followed by TMZ+ Pembrolizumab.
  * If>= 80% of contrasting enhanced tumor removed (based on T1 Post contrast magnetic resonance imaging (MRI) using cross sectional measurement), >= 7 g of tumor is resected and sufficient HSPPC-96 is generated, subjects will be included in the main cohort and will be randomized on a 1:1 basis to receive:

    * RT+TMZ +Pembrolizumab followed by TMZ+Pembrolizumab + Placebo

OR

--- RT+TMZ +Pembrolizumab followed by TMZ+Pembrolizumab+HSPPC-96

-Subjects whose tumor does not meet the criteria (unmethylated MGMT promoter and IDH wildtype by pathology) and for whom < 80 % of tumor is removed or < 7g of tumor is resected are not eligible for further intervention. Approximately 8 potentially eligible patients are screened per month, and it is anticipated that at least 1-2 per month will be accrued per site.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pre-Surgery (Step 1) Inclusion:

* Magnetic resonance imaging (MRI) findings consistent with a suspected glioblastoma (GBM) or a histologically confirmed newly diagnosed GBM that has not been treated and would benefit from further surgical resection. As vaccine needs to be generated from the patient's tumor, patients will need to be identified prior to definitive surgery.
* Preliminary assessment by the neurosurgeons that >80% of the tumor can be resected with an expectation that >7gm of tissue would be resected
* Age greater than or equal to 18 years on day of signing informed consent.
* Karnofsky performance status greater than or equal to 70.
* Tumor must be supratentorial only.
* Stereotactic biopsy will not be allowed unless there is plans for second surgery to remove greater than or equal to 80 % of the tumor.
* No prior treatment with radiation or chemotherapy for their GBM.
* No prior treatment with carmustine (Gliadel) wafers.

Post-Surgery (Step 2) Inclusion:

* Pathology must be a GBM, O6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) promoter region determined to be unmethylated and isocitrate Dehydrogenase (IDH) wild type greater than or equal to 80 % resection of contrast enhanced tumor on post operative MRI and greater than 7 grams of tumor resected are required otherwise patient is ineligible.
* Treatment must be initiated greater than or equal to 14 days and < 6 weeks from surgery.
* Craniotomy site must be adequately healed and free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of radiation. Radiation must start within 6 weeks of surgery.
* Dexamethasone dose should be less than or equal to 4 mg/day or steroid equivalent prior to starting treatment. If higher doses are needed, consult with Study Chair.
* Female subjects of childbearing potential should have a negative urine or serum pregnancy within 7 days prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required.
* Patients must have adequate organ and bone marrow function within 14 days prior to step 2 registration, as defined below:

  * Absolute neutrophil count (ANC) > 1.5 x10(9)/L; platelet count > 100 x 10(9)/L; and hemoglobin (Hb) >9.0 g/dL within 7 days prior to step 2 registration. Note: The use of transfusion or other intervention to achieve Hb greater than or equal to 9.0 g/dL is acceptable.
  * Total bilirubin < 1.5 x ULN (except in patients diagnosed with Gilbert's disease)
  * Aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT), alanine aminotransferase (ALT) serum glutamate-pyruvate transaminase (SGPT), and alkaline phosphatase (ALP) < 2.5 x ULN
  * Serum creatinine < 1.5 x ULN
  * International normalized ratio (INR), prothrombin time (PT), or activated partial thromboplastin time (APTT) as follows: In the absence of therapeutic intent to anticoagulate the patient: INR < 1.5 or PT < 1.5 x ULN or aPTT < 1.5 x ULN. In the presence of therapeutic intent to anticoagulate the patient: INR or PT and aPTT within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks before registration.
* Females of child-bearing potential (FOCBP) and males must agree to use two adequate contraception methods (give examples, e.g., hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy. Should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Male patients who father a child should notify the treating physician.

NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

1. Has not undergone a hysterectomy or bilateral oophorectomy
2. Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

   * Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.
   * Diagnosis must be made by surgical excision.
   * Patients should not be on antibiotics for any infection, but post operative antibiotics are allowed if used prophylactically but should be completed prior to starting RT.

   EXCLUSION CRITERIA:

   Pre-Surgery (Step 1) Exclusion:
   * Known history of immunodeficiency (HIV). This medical entity can be exacerbated by programmed cell death protein 1 (PD-1) blockade.
   * History of another malignancy in the previous 3 years, with a disease-free interval of < 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. Patients who have undergone a bone marrow or stem-cell transplant for any malignancy are excluded.
   * Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires chronic systemic steroids or immunosuppressive agents except as noted above. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgren's syndrome will not be excluded from the study.
   * Has a history of interstitial lung disease, non-infectious pneumonitis, or pneumonitis.
   * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Examples include:

     * Hypertension (defined as 160/95) that is not controlled on medication
     * Ongoing or active infection requiring systemic treatment
     * Symptomatic congestive heart failure
     * Unstable angina pectoris
     * Cardiac arrhythmia
     * Psychiatric illness/social situations or substance abuse disorders that would limit compliance with study requirements
     * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.
   * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
   * The effects of pembrolizumab and HSPPC-96 on the developing human fetus are unknown. For this reason and because checkpoint inhibitors and immunotherapeutic vaccines as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   * Has received prior therapy with an anti-PD-1, anti-programmed death-ligand 1 (PD-L1), anti-PD-L2, anti-4-1BB (CD137), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
   * On treatment for Hepatitis B or Hepatitis C or history of tuberculosis (TB).
   * Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Pembrolizumab are not eligible. Known hypersensitivity to any excipients of Pembrolizumab.

   Post-Surgery (Step 2) Exclusion:
   * Patients are ineligible if the tumor is not a GBM, MGMT promoter region determined to be unmethylated and IDH wild type, or if < 80 % resection of contrast enhanced tumor on post-operative MRI or < 7 grams of tumor is resected.
   * Patients who are receiving any other investigational agents.
   * Known history of immunodeficiency (HIV). This medical entity can be exacerbated by PD-1 blockade.
   * Any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment excluding steroids. Attempts should be made to have patient on lowest possible dose of steroids. These medical entities can be exacerbated by PD-1 blockade.
   * History of another malignancy in the previous 3 years, with a disease-free interval of < 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy. Patients who have undergone a bone marrow or stem-cell transplant for any malignancy are excluded.
   * Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires chronic systemic steroids or immunosuppressive agents except as noted above. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
   * Has a history of interstitial lung disease, non-infectious pneumonitis, or pneumonitis.
   * Has an active infection requiring systemic antibiotics within 10 days of surgery.
   * Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator. Examples include:

     * Hypertension (defined as 160/95) that is not controlled on medication
     * Ongoing or active infection requiring systemic treatment
     * Symptomatic congestive heart failure
     * Unstable angina pectoris
     * Cardiac arrhythmia
     * Psychiatric illness/social situations or substance abuse disorders that would limit compliance with study requirements
     * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints.
   * Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
   * The effects of pembrolizumab and HSPPC-96 on the developing human fetus are unknown. For this reason and because checkpoint inhibitors and immunotherapeutic vaccines as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
   * Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti- Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
   * On treatment for Hepatitis B or Hepatitis C or history of TB.
   * Has received a live vaccine within 30 days prior to the first dose of trial treatment
   * Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Pembrolizumab are not eligible. Known hypersensitivity to any excipients of Pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP). All collected IPD will be shared with collaborators under the terms of collaborative agreements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active. All collected individual participant data (IPD) will be available after primary analysis has been published.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0034.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Radiation therapy (RT)+Temozolomide (TZ)+Pembrolizumab+Heat Shock Protein Peptide Complex-96.(HSPPC-96). Pembrolizumab at 200mg will be administered on day 1 as a 30-minute intravenous (IV) infusion (prior to radiation therapy during RT phase) every 3 weeks on days 1, 22 and 43. Post RT, participants continue on Pembrolizumab 200mg on day 1 as a 30-minute IV infusion every 3 weeks on days 1, 22, and 43. At one year, if participants are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with HSPPC-96 vaccine if any is available. One week post RT, patients will receive weekly x 4 a dose of HSPPC-96 0.4mL intradermal vaccine. HSPPC-96 vaccine will then be given 21 days after the day 5 dose of temozolomide. HSPPC-96 vaccine will be given for 6 cycles or until supply runs out. At one year, if patients are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with HSPPC-96 if any is available. Temozolomide: TMZ will be administered on day 1 of radiation therapy (before RT treatment) and continue throughout RT at the dose of 75 mg/m^2. Post RT: The starting TMZ dose will be 150 mg/m^2/day for cycle 1, days 1-5, with a single dose escalation to 200 mg/m^2/day (days 29-33) and for all subsequent treatment if no treatment-related adverse events greater than Grade 2 are noted. TMZ will be given for 6 cycles.
- Placebo: Radiation therapy (RT)+Temozolomide (TZ)+Pembrolizumab+Placebo Vaccine. Pembrolizumab at 200mg will be administered on day 1 as a 30-minute intravenous (IV) infusion (prior to radiation therapy during RT phase) every 3 weeks on days 1, 22 and 43. Post RT, participants continue on Pembrolizumab 200mg on day 1 as a 30-minute IV infusion every 3 weeks on days 1, 22, and 43. At one year, if participants are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with placebo vaccine if any is available. One week post RT, patients will receive weekly x 4 a dose of placebo vaccine. Placebo vaccine will then be given 21 days after the day 5 dose of temozolomide. Placebo vaccine will be given for 6 cycles or until supply runs out. Participants who receive placebo will be matched for number of vaccine injections that were generated by their tumor tissue. At one year, if patients are doing well, they may continue pembrolizumab for 12 more months alone or in conjunction with placebo vaccine if any is available. Temozolomide: TMZ will be administered on day 1 of radiation therapy (before RT treatment) and continue throughout RT at the dose of 75 mg/m^2. Post RT: The starting TMZ dose will be 150 mg/m^2/day for cycle 1, days 1-5, with a single dose escalation to 200 mg/m^2/day (days 29-33) and for all subsequent treatment if no treatment-related adverse events greater than Grade 2 are noted. TMZ will be given for 6 cycles.
- Ancillary Treatment: Radiation therapy (RT) + Temozolomide (TMZ) + Pembrolizumab. Pembrolizumab at 200mg will be administered on day 1 as a 30-minute intravenous (IV) infusion (prior to radiation therapy during RT phase) every 3 weeks on days 1, 22 and 43. Post RT, participants continue on Pembrolizumab 200mg on day 1 as 30-minute IV infusion every 3 weeks on days 1, 22, and 43. After completion of 6 cycles, participants may continue on Pembrolizumab for an additional 12 months if felt to be of benefit by the treating physician. Temozolomide: TMZ will be administered on day 1 of radiation therapy (before RT treatment) and continue throughout RT at the dose of 75 mg/m^2. Post RT: The starting TMZ dose will be 150 mg/m^2/day for cycle 1, days 1-5, with a single dose escalation to 200 mg/m^2/day (days 29-33) and for all subsequent treatment if no treatment-related adverse events greater than Grade 2 are noted. TMZ will be given for 6 cycles.
- Enrolled But Not Treated: Participants were enrolled but not treated.
Period: Overall Study
Arm/Group | Vaccine | Placebo | Ancillary Treatment | Enrolled But Not Treated
Started (Tissue for vaccine production and neo-epitope monitoring.) | 8 | 9 | 15 | 58
Surgery | 8 | 9 | 15 | 56
Sufficient Vaccine Made (Minimum of Four). Participants Randomized to Arm 3 and Arm 4 (Once off treatment, continue follow-up every 8-16 weeks) | 8 | 9 | 0 | 0
No Sufficient Vaccine Made (Minimum of Four). Participants Randomized to Arm 2. (Once off treatment, continue follow-up every 8-16 weeks.) | 0 | 0 | 15 | 0
Completed | 7 | 8 | 12 | 0
Not Completed | 1 | 1 | 3 | 58
Not completed — Participants withdrew consent before surgery. | 0 | 0 | 0 | 1
Not completed — Participant withdrew consent. | 0 | 0 | 1 | 0
Not completed — Switched to alternative treatment. | 0 | 0 | 1 | 0
Not completed — Participant withdrew consent for personal reasons. | 0 | 0 | 1 | 0
Not completed — Screen failures | 0 | 0 | 0 | 51
Not completed — Chose treatment outside of UNC | 0 | 0 | 0 | 1
Not completed — Unable to comply with protocol requirements | 1 | 1 | 0 | 1
Not completed — Participant declined to participate (before treatment started) | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Ancillary Treatment | Enrolled But Not Treated | Total
Number analyzed (Participants) | 8 | 9 | 15 | 58 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 7 | 10 | 36 | 56
  >=65 years | 5 | 2 | 5 | 22 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (11.88) | 58.34 (12.6) | 58.65 (8.76) | 59.05 (14.71) | 59.9 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 6 | 29 | 38
  Male | 7 | 7 | 9 | 29 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 1 | 3
  Not Hispanic or Latino | 7 | 8 | 14 | 57 | 86
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 8 | 10
  White | 8 | 7 | 12 | 45 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 15 | 58 | 90

OUTCOME MEASURES:

1. Primary Outcome: One-year Overall Survival (OS) Rate
Description: One-year overall survival (OS) rate is defined as the percentage of participants who from time of registration survived to one year in newly diagnosed O6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) unmethylated Glioblastoma (GBM) participants treated with radiation therapy (RT) + Temozolomide (TMZ) + Pembrolizumab followed by Pembrolizumab + TMZ +/- heat-shock protein peptide complex-96 (HSPPC-96) x 6 cycles (1 cycle is 9 weeks) months. Rate of OS is measured by Kaplan-Meier method.
Time Frame: One year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 9 | 15
percentage of participants | 52.5 [24.5 to 100.0] | 71.4 [44.7 to 100.0] | 42.3 [20.4 to 87.9]

2. Secondary Outcome: Response Rate
Description: Response was determined by the Response Assessment in Neuro-Oncology Criteria (RANO) criteria and reported with 95% confidence intervals using exact binomial probability distributions. Complete response is no T1 gadolinium enhancing disease or stable or decreasing T2/fluid-attenuated inversion recovery (FLAIR). Partial response is ≥ 50% decrease in T1 gadolinium enhancing disease or stable or decreasing T2/FLAIR. Stable disease is <50% decrease but <25% increase in T1 gadolinium enhancing disease or stable or decreasing T2/FLAIR. Progressive disease is ≥25% incT1 gadolinium enhancing disease, appearance of new lesions or increase in T2/FLAIR.
Time Frame: After treatment, up to 26 months
Population: 4 out of 8 participants in vaccine group were evaluable for response. 6 out of the 9 participants in the placebo group were evaluable for response. 7 out of the 15 ancillary participants were evaluable for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 4 | 6 | 7
percentage of participants
  Complete Response | 0 [0 to 60.2] | 0 [0 to 45.9] | 0 [0 to 41.0]
  Partial Response | 0 [0 to 60.2] | 0 [0 to 45.9] | 14.3 [0.4 to 57.9]
  Stable Disease | 100.0 [39.8 to 100.] | 100.0 [54.1 to 100.0] | 28.6 [3.7 to 71.0]
  Progressive Disease | 0 [0 to 60.2] | 0 [0 to 45.9] | 57.1 [18.4 to 90.1]

3. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from registration to the time of death. Kaplan-Meier curves will be used to analyze overall survival.
Time Frame: Time from registration to the time of death or off study up to 26 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 9 | 15
Months | 14.4 [9.9 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median OS. | 14.1 [11.5 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median OS. | 10.1 [8.2 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median OS.

4. Secondary Outcome: Overall Survival at 6, 12 and 24 Months, Post-registration
Description: Participants who are alive at 6, 12 and 24 months, post-registration determined from the level of the Kaplan-Meier curves at these time points.
Time Frame: 6, 12 and 24 months, post-registration
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 9 | 15
Percentage of participants
  6 months post registration | 87.5 [67.3 to 100.0] | 100.0 [100.0 to 100.0] | 84.6 [67.1 to 100.0]
  12 months post registration | 52.5 [24.5 to 100.0] | 71.4 [44.7 to 100.0] | 42.3 [20.4 to 87.9]
  24 months post registration | 17.5 [3.0 to 100.0] | 14.3 [2.3 to 87.7] | 10.6 [1.7 to 67.1]

5. Secondary Outcome: Vaccine Cohort: Number of Adverse Events Grades 2-5, Unrelated, Unlikely, Possibly, Probably, and/or Definitely Related to Pembrolizumab
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 2 is moderate. Grade 3 is severe. Grade 4 is life-threatening. And Grade 5 is death related to adverse event.
Time Frame: Start of treatment until participant is off study, approximately 61.5 months
Measure: Number; unit: adverse events
Groups:
- Unrelated: Adverse events unrelated to Pembrolizumab.
- Unlikely Related: Adverse events unlikely related to Pembrolizumab.
- Possibly Related: Adverse events possibly related to Pembrolizumab.
- Probably Related: Adverse events probably related to Pembrolizumab.
- Definitely Related: Adverse events definitely related to Pembrolizumab.
Arm/Group | Unrelated | Unlikely Related | Possibly Related | Probably Related | Definitely Related
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
adverse events
  Grade 2 | 14 | 28 | 10 | 0 | 0
  Grade 3 | 8 | 13 | 3 | 0 | 0
  Grade 4 | 1 | 1 | 0 | 0 | 0
  Grade 5 | 1 | 0 | 0 | 0 | 0

6. Secondary Outcome: Placebo Cohort: Number of Adverse Events Grades 2-5, Unrelated, Unlikely, Possibly, Probably, and/or Definitely Related to Pembrolizumab
Description: as for outcome 5
Time Frame: Start of treatment until participant is off study, approximately 61.5 months
Measure: Number; unit: Adverse events
Arm/Group | Unrelated | Unlikely Related | Possibly Related | Probably Related | Definitely Related
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9
Adverse events
  Grade 2 | 5 | 19 | 11 | 4 | 2
  Grade 3 | 8 | 5 | 1 | 7 | 1
  Grade 4 | 0 | 0 | 0 | 1 | 1
  Grade 5 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Ancillary Treatment Cohort: Number of Adverse Events Grades 2-5, Unrelated, Unlikely, Possibly, Probably, and/or Definitely Related to Pembrolizumab
Description: as for outcome 5
Time Frame: Start of treatment until participant is off study, approximately 61.5 months
Measure: Number; unit: Adverse Events
Arm/Group | Unrelated | Unlikely Related | Possibly Related | Probably Related | Definitely Related
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 15
Adverse Events
  Grade 2 | 17 | 43 | 13 | 0 | 2
  Grade 3 | 18 | 25 | 7 | 3 | 2
  Grade 4 | 1 | 5 | 2 | 0 | 1
  Grade 5 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Mean Symptom Severity Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT).
Description: To evaluate the occurrence of symptoms and correlate to disease progression and tolerance to treatment using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT). Participants rate their symptoms on a questionnaire using an 11-point scale (0-10). 0 is "not present" and 10 is "as bad as you can imagine." Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity measures. Higher score indicates worse severity.
Time Frame: Baseline, end of treatment or discontinuation, and 30 days after last dose
Population: There are different numbers for overall participants analyzed because we don't have that data available (i.e., a few participants didn't do a baseline questionnaire).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 8 | 13
Score on a scale
  Baseline | 1.4 (0.8) | 1.3 (0.9) | 1.2 (1.1)
  End of treatment or discontinuation: number analyzed (Participants) | 2 | 6 | 6
  End of treatment or discontinuation | 4.0 (1.5) | 1.4 (0.8) | 2.4 (1.8)
  30 days after last dose: number analyzed (Participants) | 0 | 1 | 3
  30 days after last dose |  | 1.7 | 1.9 (0.5)

9. Secondary Outcome: Mean Symptom Interference Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT).
Description: To evaluate the occurrence of symptoms and correlate to disease progression and tolerance to treatment using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT). Participants rate their symptoms on a questionnaire using an 11-point scale (0-10) of how much symptoms interfered with different aspects of a patient's life in the last 24 hours such as general activity, mood, work, relations with other people, walking and enjoyment of life. 0 is "not present" and 10 is "as bad as you can imagine." Differences of at least 2 points will be classified as the minimum clinically meaningful change in the symptom severity measures.
Time Frame: Baseline, end of treatment or discontinuation, and 30 days after last dose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 8 | 13
Score on a scale
  Baseline | 2.9 (2.4) | 1.9 (1.4) | 2.2 (2.7)
  End of treatment or discontinuation: number analyzed (Participants) | 2 | 6 | 6
  End of treatment or discontinuation | 7.0 (4.0) | 1.6 (2.8) | 4.3 (4.1)
  30 days after last dose: number analyzed (Participants) | 0 | 1 | 3
  30 days after last dose |  | 6.0 | 3.1 (2.9)

10. Secondary Outcome: Percentage of Participants Rating Their Symptom Severity to Be 5 or Greater (on a 0-10) Scale Using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT)
Description: Percentage of participants rating their symptom severity to be 5 or greater (on a 0-10) scale using the MD Anderson Symptom Inventory-Brain Tumor Module (MDASI-BT). Participants rate their symptoms on a questionnaire using an 11-point scale (0-10). 0 is "not present" and 10 is "as bad as you can imagine."
Time Frame: Baseline, end of treatment or discontinuation, and 30 days after last dose
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 8 | 13
Percentage of participants
  Baseline | 38 [9 to 76] | 63 [25 to 92] | 54 [25 to 81]
  End of treatment or discontinuation: number analyzed (Participants) | 2 | 6 | 6
  End of treatment or discontinuation | 83 [36 to 100] | 100 [16 to 100] | 83 [36 to 100]
  30 days after last dose: number analyzed (Participants) | 0 | 1 | 3
  30 days after last dose |  | 100 [29 to 100] | 100 [3 to 100]

11. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from registration to the time of confirmed progression. Progression was measured by the immunotherapy response assessment for neuro-oncology (iRANO) criteria. Progressive disease is ≥25% increase in the sum of bi-perpendicular diameters of enhancing disease or new lesions or significant worsened T2/fluid-attenuated inversion recovery (FLAIR) or significant clinical decline.
Time Frame: Time from registration to the time of confirmed progression, an average of 9 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vaccine | Placebo | Ancillary Treatment
Number analyzed (Participants) | 8 | 9 | 15
Months | 13.7 [9.92 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median PFS. | 8.0 [5.94 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median PFS. | 10.3 [5.9 to NA] — The follow-up is not long enough to estimate the upper bound of the confidence intervals for median PFS.

12. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 61.5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo | Ancillary Treatment | Enrolled But Not Treated
Number analyzed (Participants) | 8 | 9 | 15 | 58
Participants | 8 | 9 | 15 | 2

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 61.5 months.
Arm/Group | Vaccine | Placebo | Ancillary Treatment | Enrolled But Not Treated
All-Cause Mortality (participants affected / at risk) | 6/8 | 4/9 | 10/15 | 0/58
Serious Adverse Events (participants affected / at risk) | 6/8 | 4/9 | 8/15 | 2/58
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 12/15 | 2/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=8) | Placebo (N=9) | Ancillary Treatment (N=15) | Enrolled But Not Treated (N=58)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema cerebral (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, altered mental status (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=8) | Placebo (N=9) | Ancillary Treatment (N=15) | Enrolled But Not Treated (N=58)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (5) | 6 (14) | 5 (20) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (13) | 2 (4) | 3 (21) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 5 (8) | 5 (12) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (2) | 1 (3) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders - Other, Hearing Loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Endocrine disorders - Other, Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, Eye Pressure (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, left eye rotating lateral side (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye disorders - Other, left eyelid droop (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (9) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (5) | 3 (4) | 8 (10) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (5) | 2 (9) | 2 (4) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (6) | 1 (2) | 2 (8) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 2 (2) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 3 (3) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (12) | 2 (5) | 3 (6) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (12) | 1 (1) | 1 (1) | 0 (0)
Left ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (41) | 3 (32) | 3 (32) | 2 (5)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Bilateral Lower Extremity Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Bilateral Shin Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Phantosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, left hand numbness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, left hemineglect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 2 (7) | 2 (6) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (18) | 3 (7) | 4 (15) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary infiltrate (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, kidney stones (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, polydypsia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (6) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Increased Facial Hair (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Oral Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, psoriasis(flare) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Head pain (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaccination site lymphadenopathy (General disorders) | 1 (10) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision decreased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Weight gain (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (10) | 2 (14) | 2 (17) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT03018288/Prot_SAP_003.pdf
  • Informed Consent Form (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT03018288/ICF_001.pdf